CLINICAL TRIAL: NCT04535063
Title: Convalescent Plasma as Potential Therapy for Severe COVID-19 Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno (Other)
Responsible Party: Principal Investigator, Ricardo Valentini, Medical Doctor, Centro de Educación Medica e Investigaciones Clínicas Norberto Quirno
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RValentini
Record Dates: First submitted 2020-08-29; First posted 2020-09-01 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Covid19 Pneumonia

STUDY DESIGN:
Intervention Model Description: patients with severe COVID19 pneumonia will be recruited to a single arm therapy group with convalescent plasma from recovered patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- severe pneumonia arm (Other): patients with severe COVID19 pneumonia defined by: spontaneous breathing patients with respiratory failure requiring O2 nasal cannula more than 3 L/min or reservoir oxygen mask and SaO2 less than 95% or patients with critical pneumonia define by mechanical ventilation with less than 300 mmHg PaO2/FiO2 or shock or multi-organic dysfunction
  Interventions: Biological: COVID19 convalescent plasma infusion

INTERVENTIONS:
Biological: COVID19 convalescent plasma infusion — intravenous infusion of 300-600 mL of convalescent plasma with an antibody title more than 3 according to chemiluminescent microparticle immunoassay (Architect Plus Abbott)

SUMMARY:
To determinate feasibility, safety and outcome with convalescent plasma in patients with severe COVID-19 penumonia

DETAILED DESCRIPTION:
COVID-19 convalescent plasma will be infused to patients with severe COVID-19 pneumonia to determine feasibility, safety and clinical outcome efficacy by survival at-28 days. Data will be compared with match control arm patients without plasma infusion

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18, and non-pregnant women
* Severe or critical COVID-19 disease define by one or more of the following: blood oxygen saturation ≤ 94% on supplemental oxygen by nasal cannula at least 3 L/min, non-rebreathing mask (NRO2-mask) or on noninvasive ventilation; and pulmonary infiltrates with >50% increase within 24 to 48 hours in chest-X-ray or chest CT. Life-threatening disease was defined as one or more of the following: respiratory failure on mechanical ventilation with PaO2 / FiO2 less than 300 mm Hg, septic shock, and/or multiple organ dysfunction.

  * 10 days from the onset of symptoms or ≤ 7 days on mechanical ventilation. -

Exclusion Criteria:

* More than 10 days from symptoms onset or more than 7 days on mechanical ventilation
* Pregnancy
* Contraindication for plasma infusion because anaphylaxis history
* Patients with high risk of circulatory overload
* Limitation of therapeutic efforts
* Refractory shock define by norepinephrine dose more than 1 ug/k/min
* SOFA score more than 15 points at the moment of the protocol inclusion i Coagulopathy with requirements of plasma infusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-04-18 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
28 days survival | 28 days
  number of subjects surviving at 28 days from plasma infusion

SECONDARY OUTCOMES:
efficacy of plasma infusion according to antibodies levels in the infuse bags | 28 days
  comparison of clinical efficacy according antibodies levels
clinical efficacy of plasma infusion according to frame time from symptoms onset and hospitalization | 28 days
  we will search if clinical efficacy is better when the earlier the infusion is decided
change in clinical WHO ordinal scale from 1 to 10 points | 14 days
  WHO clinical scale is a measure of patient progression through the health-care system with 1 point asymptomatic patient and 10 patient dead

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Educación Médica e Investigaciones Clínicas, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No
we will to share results to compare data with other studies with convalescent plasma infusion in COVID 19 patients after finishing our study